CLINICAL TRIAL: NCT06448676
Title: Head-to-Head Comparison of the Efficacy and Safety of All Five Commercially Available Botulinum Neurotoxin Type A Products for the Treatment of Glabellar Rhytides: A Multicenter, Triple-Blind, Randomized Controlled Trial
Brief Title: Head-to-Head Comparison of All Botulinum Neurotoxin Type A Products for Glabellar Rhytides
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: Universitair Medical Centrum Groningen (Unknown)
Responsible Party: Principal Investigator, Prof. dr. J. de Lange, MD DMD, Prof. dr. Jan de Lange, MD DMD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-514936-26-00
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Wrinkle
MeSH Terms: interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: This study is a triple-blind, multi-center, parallel-group randomized controlled trial designed to compare the efficacy and safety of onabotulinumtoxinA, abobotulinumtoxinA, incobotulinumtoxinA, prabotulinumtoxinA, and daxibotulinumtoxinA, for the treatment of glabellar rhytides.
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Trial participants, data collectors, the statistician, and outcome assessors were blinded to the study-group assignments. Blinded syringes are labeled a sticker containing no information other than the allocated study number. After reconstitution, syringes were stored under hygienic non-sterile conditions between 39-46F in medical refrigerators. The safety related to this sterile transfer is substantiated by several studies.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (7):
- OnabotulinumtoxinA: 20 units (Active Comparator): 20 units (4-4-4-4-4) Commercial Name: Botox® Producing Company: Allergan, an AbbVie company Location: Dublin, Ireland Additional Commercial Names: Vistabel® (in some regions, especially Europe)
  Interventions: Drug: Botulinum toxin type A
- IncobotulinumtoxinA: 20 units (Active Comparator): 20 units (4-4-4-4-4) Commercial Name: Xeomin® Producing Company: Merz Pharmaceuticals Location: Frankfurt, Germany Additional Commercial Names: Bocouture® (for aesthetic use in some regions)
  Interventions: Drug: Botulinum toxin type A
- AbobotulinumtoxinA: 50 (Speywood) units (Active Comparator): 50 units (10-10-10-10-10) Commercial Name: Dysport® Producing Company: Ipsen Biopharmaceuticals, Inc. Location: Paris, France Additional Commercial Names: Azzalure® (for aesthetic use in some regions)
  Interventions: Drug: Botulinum toxin type A
- AbobotulinumtoxinA: 60 (Speywood) units (Active Comparator): 60 units (12-12-12-12-12) Commercial Name: Dysport® Producing Company: Ipsen Biopharmaceuticals, Inc. Location: Paris, France Additional Commercial Names: Azzalure® (for aesthetic use in some regions)
  Interventions: Drug: Botulinum toxin type A
- PrabotulinumtoxinA 20 units (Active Comparator): 20 units (4-4-4-4-4) Commercial Name: Jeuveau® Producing Company: Evolus, Inc. Location: Newport Beach, California, USA Additional Commercial Names: Nuceiva® (for aesthetic use in some regions)
  Interventions: Drug: Botulinum toxin type A
- Excluded: DaxibotulinumtoxinA 20 units (reason for exclusion: not available in the EU) (Active Comparator): 20 units (4-4-4-4-4) Commercial Name: Daxxify® Producing Company: Revance Therapeutics, Inc. Location: Nashville, Tennessee, USA
  Interventions: Drug: Botulinum toxin type A
- Excluded: LetibotulinumtoxinA-wlbg: 20 units (reason for exclusion: not available in the EU). (Active Comparator): Arm Description: 20 units (4-4-4-4-4) Commercial Name: Letybo® Producing Company: Hugel Inc. Location: Chuncheon-si, South Korea
  Interventions: Drug: Botulinum toxin type A

INTERVENTIONS:
Drug: Botulinum toxin type A — Head-to-head comparison of all commercially available botulinum neurotoxin type A products

SUMMARY:
Study Type: This is a multicenter, triple-blind, randomized controlled trial.

Purpose: The goal of this clinical trial is to compare the effectiveness and safety of all five commercially available Botulinum Neurotoxin Type A (BoNT-A) products for treating glabellar rhytides, commonly known as frown lines. This study is designed to provide comprehensive data on how these treatments compare in terms of improving frown lines and the duration of their effects.

Main Questions the Study Aims to Answer:

Which BoNT-A product provides the longest lasting effect on reducing glabellar rhytides? How do these products compare in terms of safety and the occurrence of side effects?

Participant Tasks:

Women aged 18 years or older with moderate to severe glabellar lines will participate.

Participants will receive injections of a BoNT-A product into specific facial muscles.

They will need to take weekly photographs using their smartphones to document changes in their frown lines.

These photos will be securely sent to our research team for analysis. Participants will complete questionnaires at the start and end of the study to assess their satisfaction, quality of life, and any changes in their condition.

Comparison Group:

Researchers will compare participants receiving different types of BoNT-A products to see which one is more effective at reducing frown lines and maintaining these effects over time.

The safety profiles of these products will also be compared to determine which has the fewest and least severe side effects.

This study aims to fill important gaps in our understanding of Botulinum Neurotoxin Type A treatments, guiding more effective clinical decisions and improving patient outcomes.

DETAILED DESCRIPTION:
Background: Glabellar rhytides, commonly known as frown lines, are a significant aesthetic concern for many individuals, leading to increasing utilization of Botulinum Neurotoxin Type A (BoNT-A) treatments. Despite multiple products being available, comprehensive comparative data on their efficacy and safety are limited. This trial aims to fill this evidence gap by evaluating and comparing the effectiveness and safety profiles of all five FDA-approved BoNT-A products.

Methods: Conducted across several clinical sites, this multicenter, triple-blind, randomized controlled trial will involve a structured intervention where participants receive one of five different BoNT-A formulations. The study employs a stringent blinding and randomization process to ensure the objectivity and reliability of the results. Data on treatment efficacy, safety, and participant-reported outcomes will be collected at baseline and follow-up through direct clinical assessments and secure digital communication methods.

Data Collection and Analysis: Data collection will include baseline and 16-week follow-up assessments using standardized clinical scales and self-reported question anaires. Participants will document 30 weekly progress through standardized 'selfie' photos using a secure, encrypted application to ensure data privacy. The primary outcome, the duration of treatment efficacy, will be analyzed using Kaplan-Meier survival analysis. Secondary outcomes, including the incidence of adverse events and participant satisfaction, will be analyzed using repeated measures ANOVA and logistic regression. Detailed duration of effect will be assessed using Kaplan-Meier curves and Cox proportional hazards models.

Statistical Analysis: The study is powered to detect meaningful clinical differences between the treatment groups with a high degree of statistical confidence. The analysis will explore treatment effects over time and assess factors influencing treatment efficacy and safety.

Conclusion: By rigorously comparing all available BoNT-A products, this study will provide critical insights into their relative effectiveness and safety, significantly informing clinical decision-making and optimizing patient care strategies for treating glabellar lines. The findings are expected to enhance the understanding of treatment dynamics and guide future therapeutic approaches in aesthetic medicine.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18 years or over, with moderate to severe glabellar lines
* Willing to provide written informed consent
* American Society of Anesthesiologists (ASA) Physical Status Classification 1 or 2

Exclusion Criteria:

* ASA Classification 3 or over
* History of hypersensitivity or adverse reactions to botulinum toxin or any of its components
* Infection at the injection site
* Previous treatment with botulinum toxin (lifetime)
* Pregnant or breastfeeding women
* Neuromuscular disorders or conditions that could interfere with the study assessments

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-10-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Duration of Clinical Efficacy | From baseline to week 16
  Period until loss of treatment effect, measured as the percentage of participants who maintain at least a 1-point improvement in glabellar line severity at maximum frown from baseline to week 16, assessed using the "four-point clinical severity score for glabellar frown lines" developed by Honeck.

SECONDARY OUTCOMES:
Duration of Clinical Efficacy | Kaplan-Meier survival curves and Cox proportional hazards models to analyze the time to complete loss of effect across the entire study duration (From baseline to week 30)
  Median time to loss of effect
Incidence of Adverse Events (AEs) | From baseline to week 16
  Occurrences of adverse events such as ptosis, strabismus, and eyelid sensory disorders throughout the study period
Quality of Life (FACE-Q) | From baseline to week 16
  FACE-Q Psychological Wellbeing Scores, (values 10-40), higher score means a better outcome
Social Functioning (FACE-Q) | From baseline to week 16
  FACE-Q Social Scores, (values 8-32), higher score means a better outcome
Satisfaction with the Result (FACE-Q) | From baseline to week 16
  FACE-Q Outcome Scores, (values 6-24), higher score means a better outcome
Depressive Symptoms | Baseline to week 4
  Hospital Anxiety and Depression Scale (HADS) Depression Scores, (values 0-21), higher score means a worse outcome
Anxiety Symptoms | Baseline to week 4
  Hospital Anxiety and Depression Scale (HADS) Anxiety Scores, (values 0-21), higher score means a worse outcome
Migraine Symptoms | Baseline to week 4
  Migraine Disability Assessment (MIDAS) Scores, (values 0-21+), higher score means a worse outcome
Headache Symptoms | Baseline to week 4
  Headache Impact Test (HIT-6) Scores, (values 36-78), higher score means a worse outcome
Side Effects (FACE-Q) | First 2 weeks after treatment
  FACE-Q Early Life Impact Scores, (values 17-68), higher score means a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Jan de Lange, MD DMD PhD, Principal Investigator — Amsterdam University Medical Centers

REFERENCES:
- [Background] Decates T, de Wijs L, Nijsten T, Velthuis P. Numbers on injectable treatments in the Netherlands in 2016. J Eur Acad Dermatol Venereol. 2018 Aug;32(8):e328-e330. doi: 10.1111/jdv.14877. Epub 2018 Mar 6. No abstract available. PMID 29444367
- [Background] Decates TS, Velthuis P, Zarringam D, Bruin L, Schepers RH, van der Lei B. Upward trend in number of injectable treatments in the Netherlands 2016-2019. J Cosmet Dermatol. 2021 Sep;20(9):3049-3051. doi: 10.1111/jocd.14339. Epub 2021 Jul 19. No abstract available. PMID 34403196
- [Background] Steenen SA, Bauland CG, de Lange J, van der Lei B. Complications After Botulinum Neurotoxin Type A and Dermal Filler Injections: Data From a Large Retrospective Cohort Study. Aesthet Surg J. 2023 Jan 9;43(1):NP56-NP63. doi: 10.1093/asj/sjac228. No abstract available. PMID 35953448
- [Background] Jia Z, Lu H, Yang X, Jin X, Wu R, Zhao J, Chen L, Qi Z. Adverse Events of Botulinum Toxin Type A in Facial Rejuvenation: A Systematic Review and Meta-Analysis. Aesthetic Plast Surg. 2016 Oct;40(5):769-77. doi: 10.1007/s00266-016-0682-1. Epub 2016 Aug 5. PMID 27495260
- [Background] Zargaran D, Zoller FE, Zargaran A, Mosahebi A. Complications of facial cosmetic botulinum toxin A injection: analysis of the UK Medicines & Healthcare Products Regulatory Agency registry and literature review. J Plast Reconstr Aesthet Surg. 2022 Jan;75(1):392-401. doi: 10.1016/j.bjps.2021.05.074. Epub 2021 Jun 17. PMID 34456155
- [Background] Gostimir M, Liou V, Yoon MK. Safety of Botulinum Toxin A Injections for Facial Rejuvenation: A Meta-Analysis of 9,669 Patients. Ophthalmic Plast Reconstr Surg. 2023 Jan-Feb 01;39(1):13-25. doi: 10.1097/IOP.0000000000002169. Epub 2022 Mar 30. PMID 35353777
- [Background] Zargaran D, Zoller F, Zargaran A, Rahman E, Woollard A, Weyrich T, Mosahebi A. Complications of Cosmetic Botulinum Toxin A Injections to the Upper Face: A Systematic Review and Meta-Analysis. Aesthet Surg J. 2022 Apr 12;42(5):NP327-NP336. doi: 10.1093/asj/sjac036. PMID 35178552
- [Background] Li X, Sui C, Xia X, Chen X. Efficacy and Safety of Botulinum Toxin Type A for Treatment of Glabellar Lines: A Network Meta-Analysis of Randomized Controlled Trials. Aesthetic Plast Surg. 2023 Feb;47(1):365-377. doi: 10.1007/s00266-022-03018-y. Epub 2022 Sep 12. PMID 36097079
- [Background] Kerscher M, Fabi S, Fischer T, Gold M, Joseph J, Prager W, Rzany B, Yoelin S, Roll S, Klein G, Maas C. IncobotulinumtoxinA Demonstrates Safety and Prolonged Duration of Effect in a Dose-Ranging Study for Glabellar Lines. J Drugs Dermatol. 2021 Oct 1;20(10):1052-1060. doi: 10.36849/JDD.6377. PMID 34636520
- [Background] Polacco MA, Singleton AE, Barnes CH, Maas C, Maas CS. A Double-Blind, Randomized Clinical Trial to Determine Effects of Increasing Doses and Dose-Response Relationship of IncobotulinumtoxinA in the Treatment of Glabellar Rhytids. Aesthet Surg J. 2021 May 18;41(6):NP500-NP511. doi: 10.1093/asj/sjaa220. PMID 32722793
- [Background] Joseph J, Moradi A, Lorenc ZP, Coleman K, Ablon G, Kaufman-Janette J, Cox SE, Campbell A, Dayan S, Berg AK, Munavalli G. AbobotulinumtoxinA for the Treatment of Moderate-to-Severe Glabellar Lines: A Randomized, Dose-Escalating, Double-Blind Study. J Drugs Dermatol. 2021 Sep 1;20(9):980-987. doi: 10.36849/jdd.6263. PMID 34491016
- [Background] Lorenc ZP, Adelglass JM, Avelar RL, Baumann L, Beer KR, Cohen JL, Cox SE, Dayan SH, Dover JS, Downie JB, Draelos ZD, Goldman MP, Gross JE, Joseph JH, Kaufman-Janette J, Moy RL, Nestor M, Schlessinger J, Smith SR, Weiss RA. The Second of Two One-Year, Multicenter, Open-Label, Repeat-Dose, Phase II Safety Studies of PrabotulinumtoxinA for the Treatment of Moderate to Severe Glabellar Lines in Adult Patients. Aesthet Surg J. 2021 Nov 12;41(12):1423-1438. doi: 10.1093/asj/sjaa382. PMID 33944913
- [Background] Taylor SC, Grimes PE, Joseph JH, Jonker A, Avelar RL. PrabotulinumtoxinA for the Treatment of Moderate-to-Severe Glabellar Lines in Adult Patients With Skin of Color: Post Hoc Analyses of the US Phase III Clinical Study Data. Dermatol Surg. 2021 Apr 1;47(4):516-521. doi: 10.1097/DSS.0000000000002864. PMID 33165078
- [Background] Dayan S, Joseph J, Moradi A, Lorenc ZP, Coleman K, Ablon G, Kaufman-Janette J, Cox SE, Campbell A, Munavalli G, Prygova I. Subject satisfaction and psychological well-being with escalating abobotulinumtoxinA injection dose for the treatment of moderate to severe glabellar lines. J Cosmet Dermatol. 2022 Jun;21(6):2407-2416. doi: 10.1111/jocd.14906. Epub 2022 Apr 12. PMID 35266281
- [Background] Bertucci V, Solish N, Kaufman-Janette J, Yoelin S, Shamban A, Schlessinger J, Snyder D, Gallagher C, Liu Y, Shears G, Rubio RG. DaxibotulinumtoxinA for Injection has a prolonged duration of response in the treatment of glabellar lines: Pooled data from two multicenter, randomized, double-blind, placebo-controlled, phase 3 studies (SAKURA 1 and SAKURA 2). J Am Acad Dermatol. 2020 Apr;82(4):838-845. doi: 10.1016/j.jaad.2019.06.1313. Epub 2019 Nov 29. PMID 31791824
- [Background] Steenen SA, Bauland CG, van der Lei B, Su N, van Engelen MDG, Anandbahadoer-Sitaldin RDRRAL, Koeiman W, Jawidan T, Hamraz Y, Lange J. Head-to-head comparison of 4 hyaluronic acid dermal fillers for lip augmentation: A multicenter randomized, quadruple-blind, controlled clinical trial. J Am Acad Dermatol. 2023 Apr;88(4):932-935. doi: 10.1016/j.jaad.2022.11.012. Epub 2022 Nov 9. No abstract available. PMID 36370906
- [Background] Shome D, Kapoor R, Khare S. Two different types of botulinum toxins: Is there a difference in efficacy and longevity? J Cosmet Dermatol. 2019 Dec;18(6):1635-1641. doi: 10.1111/jocd.12949. Epub 2019 May 28. PMID 31135088
- [Background] Bohart Z, Dashtipour K, Kim H, Schwartz M, Zuzek A, Singh R, Nelson M. Real-world differences in dosing and clinical utilization of OnabotulinumtoxinA and AbobotulinumtoxinA in the treatment of upper limb spasticity. Toxicon. 2024 Apr;241:107678. doi: 10.1016/j.toxicon.2024.107678. Epub 2024 Mar 4. PMID 38447766
- [Background] Honeck P, Weiss C, Sterry W, Rzany B; Gladys study group. Reproducibility of a four-point clinical severity score for glabellar frown lines. Br J Dermatol. 2003 Aug;149(2):306-10. doi: 10.1046/j.1365-2133.2003.05436.x. PMID 12932236